CLINICAL TRIAL: NCT05836961
Title: Evaluating Effectiveness of Benazir Nashonuma Program (BNP) on Maternal and Infant Outcomes: A Non-randomized Intervention Study in Sindh and Punjab
Brief Title: Impact of Benazir Nashonuma Program (BNP) on Maternal and Child Nutritional Status
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: International Food Policy Research Institute (Other); Bill and Melinda Gates Foundation (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguished University Professor and Founding Director of the Institute for Global Health and Development and the Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNP Study
Record Dates: First submitted 2023-03-13; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-01

CONDITIONS: Low Birthweight; Stunting; Wasting; Malnutrition, Child; Iron Deficiency Anemia; Dietary Habits
Keywords: Intervention study; Maternal and child nutrition; Benazir Nashonuma Program (BNP); Low birthweight; Stunting
MeSH Terms: conditions — Growth Disorders; Cachexia; Child Nutrition Disorders; Anemia, Iron-Deficiency; Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BNP enrolled (Experimental): Pregnant women in their first or second trimester who have been enrolled in BNP
  Interventions: Other: Benazir Nashonuma Program (BNP)
- BNP non-enrolled (No Intervention): Pregnant women in their first or second trimester who are not enrolled in BNP

INTERVENTIONS:
Other: Benazir Nashonuma Program (BNP) — Dietary supplement for pregnant women and lactating mothers during the first six months of lactation:
  Maamta is a 75-gram sachet made from peanut butter with 400 kcal of energy
  Dietary supplement for children aged 6-23 months:
  Wawamum is a lipid-based nutrient supplement consisting of skimmed milk powder, micronutrients, vegetable oil, roasted chickpeas and antioxidants. Wawamum covers the recommended daily dose of most micronutrients and 255 kcal of energy (1/4 of daily energy requirements for children in this age range)
  Conditional Cash Transfers (CCT):
  This includes stipends of PKR 2000 during pregnancy contingent on three antenatal care visits, consuming SNF, attending awareness sessions on health and nutrition, getting two doses of tetanus toxoid and institutional delivery. After delivery PKR 2000/- for boys and 2500/- for girls are paid as incentives conditioned on getting child's birth registered, routine immunization and consumption of SNF by the child from 6-23 months
  Arms: BNP enrolled

SUMMARY:
The purpose of this study is to evaluate the impact of Benazir Nashonuma Program (BNP) which includes specialized nutritious food (SNF) augmented with specific reproductive health interventions during pregnancy on proportion of low birthweight babies and stunting among children, in low income setting of Pakistan. The study aims to answer if:

1. Utilization of Benazir Nashonuma Program (BNP) among pregnant women is effective in reducing the proportion of low birthweight babies, compared to pregnant women who are not utilizing the program, among low income setting population.
2. Utilization of Benazir Nashonuma Program (BNP) is effective in reducing the proportion of stunting among children, compared to those not utilizing the program, among low income setting population.

Participants who are enrolled in the Benazir Nashonuma Program (receiving intervention) and those who are not enrolled (not receiving intervention) will be followed throughout pregnancy till delivery. After delivery mother-baby dyad will be followed for a period of 12 months. Compliance of supplementation will be measured, and outcomes (low birthweight and stunting) observed throughout the follow up.

DETAILED DESCRIPTION:
Malnutrition in Pakistan is a major and pervasive public health issue. Every four under five children in our country are reported to be stunted, with a mighty prevalence of 40.2% stunting as reported in the National Nutritional Survey of Pakistan 2018. Pakistan also shares one of the highest burden of low birthweight (LBW) where 19% babies in urban and 32% in rural are born with weight <2500 grams. LBW babies have a higher risk of death compared to full term babies and contributes to 60-80% of all neonatal deaths.

The first 1000 days of life, the time from conception to 2 years of age, is a critical period, providing a window of opportunity for interventions to improve maternal and child nutrition and health outcomes including stunting and other nutritional markers. Availability and access to primary healthcare and nutrition services during pregnancy and the first two years of life can help prevent undernutrition and reduce infections in early life, helping reduce maternal and infant mortality, and preventing the lifelong and intergenerational consequences of malnutrition. Evidence-based nutrition interventions, especially the combination of BEP and small quantity lipid nutrient supplements have been shown to be effective in improving birth outcomes and reducing child stunting.

BNP is a health and nutrition CCT programme, with the aim to address stunting in children under 23 months of age. The CCT and Specialized Nutritious Food (SNF) are provided to Benazir Income Support Programme (BISP) participating women during pregnancy and lactation up to 6 months and to children aged 6-23 months contingent on their participation in and adherence to BNP interventions. In addition to the programme components, the pre-existing standard of care interventions including antenatal and postnatal care, childhood immunizations, growth monitoring and behavior change communication (BCC) activities, i.e., awareness sessions on health, nutrition and hygiene.

The primary study objectives are to assess the impact of intervention (BNP) on:

* Proportion of babies born with low birthweight.
* Prevalence of stunting among infants at 6 and 12 months of age

The secondary objectives related to maternal outcomes are to assess the impact of intervention on:

* Dietary diversity of women
* Mean nutrient intake including energy in kilo calories.
* Prevalence of iron deficiency anemia among lactating women.
* Proportion of pregnant women using reproductive health services.

The secondary objectives related to newborn and infant outcomes are to assess the impact of the intervention on:

* Prevalence of wasting among infants at 6 and 12 months of age.
* Incidence of anemia among infants at 6- and 12-months of age
* Infant and child feeding practices among infants at 6 and 12 months of age.
* Neurodevelopmental outcomes (cognitive, language and motor development) using Bayley Scales of Infant and Toddler Development (BSID-IV) at 6 months, and 12 months of age among children.

Other objectives include following:

* To measure receipt and utilization of BEP supplementation among pregnant and lactating women enrolled in BNP.
* To measure receipt and utilization on BEP supplementation among children under 12 months of age enrolled in BNP
* Household food insecurity status (using the Food Insecurity Experience Scale).

ELIGIBILITY:
Inclusion Criteria:

Intervention arm: All pregnant women in their first or second trimester, who are enrolled in Benazir Nashonuma Program (BNP).

Non-intervention arm: All pregnant women in their first or second trimester, who are not enrolled in Benazir Nashonuma Program (BNP).

Exclusion Criteria:

* Women who intend to migrate or relocate for more than 3 months during the study period will be excluded from the study.
* Women in the non intervention group who are consuming specialized nutritious food (SNF) from any source at the time of enrollment will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of low birthweight | Within 48-hours of delivery
  Birth weight of less than 2500 g (up to and including 2499 g) within 48 hours of delivery
Prevalence of stunting | At 6 months of age
  Height-for-age ≤-2 SD of the WHO Child growth standards median
Prevalence of stunting | At 12 months of age
  Height-for-age ≤-2 SD of the WHO Child growth standards median

SECONDARY OUTCOMES:
Prevalence of wasting | At 6 and 12 months of age
  Weight-for-height ≤-2 SD of the WHO Child growth standards median.
Prevalence of Iron deficiency anemia in pregnant women | At 9th month on pregnancy
  Hemoglobin levels below 11 g/dl, serum ferritin less than or equal to 30 ng/ml, mean corpuscular volume MCV below 95 fl will be considered diagnostic of iron deficiency anemia
Prevalence of Iron deficiency anemia in infants | 2 point times: At 6 and 12 months of age
  Hemoglobin concentration of less than 11.0 g/dl and ferritin levels of less than 15 micrograms/L
Number of antenatal care (ANC) visits during pregnancy | At delivery
  Attending at least 8 ANC consultations in a health facility/clinic
Number of women who had an Institutional delivery | At delivery
  Having delivered in a health facility
Number of women who had Skilled birth attendance | At delivery
  Birth attended by a skilled health personnel
Number of women who had Postnatal care (PNC) check ups | 3 months after delivery
  Receiving a postnatal health check while in a facility or at home within 6-weeks of postnatal period
Mean nutrient intake of energy in kilocalories of the pregnant woman | At 9th month of pregnancy
  Mean nutrient intake of energy in kilocalories using 24-hour recall.
Prevalence of infants who were ever breastfed | At 12 months of age
  Number of infants who were breastfed at least once
Prevalence of infants who had early initiation of breastfeeding | At 12 months of age
  Number of infants who were put to the breast within one hour of birth
Prevalence of infants who were exclusively breastfed | At 12 months of age
  Number of of infants aged 0-5 months who were fed exclusively with breast milk during the previous day
Prevalence of infants who consumed a minimum acceptable diet | At 12 months of age
  Number of infants 6-12 months of age who consumed a minimum acceptable diet during the previous day
Prevalence of infants with minimum dietary diversity | At 12 months of age
  Number of infants 6-12 months of age who consumed foods and beverages from at least four out of eight defined food groups during the previous day
Mean scores of Neurodevelopmental outcomes of the infant | At 12 months of age
  Neurodevelopmental outcomes of the children will be assessed using Bayley Scales of Infant and Toddler Development (BSID-IV). Mean scores will be reported for cognitive, language and motor development of the infant using Bayley's scales. Higher scores in the Bayley Scales indicate better outcomes
Number of women consuming specialized nutritious food (SNF) | At 6 months after delivery
  Utilization of supplementation (SNF) by the woman during pregnancy and first 6 months of lactation after delivery
Number of infants consuming specialized nutritious food (SNF) | At 12 months of age
  Utilization of supplementation (SNF) by the infant from 6-23 months of age

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan Office, Dadu, Sindh, Pakistan